CLINICAL TRIAL: NCT00499369
Title: Phase III Trial of Irinotecan-Based Chemotherapy Plus Cetuximab (NSC-714692) or Bevacizumab (NSC-704865) as Second-Line Therapy for Patients With Metastatic Colorectal Cancer Who Have Progressed on Bevacizumab With Either FOLFOX, OPTIMOX or XELOX
Brief Title: Irinotecan and Cetuximab With or Without Bevacizumab in Treating Patients With Metastatic Colorectal Cancer That Progressed During First-Line Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to inadequate accrual, study was terminated and limited outcome data was reported.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00784; NCI-2009-00784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-SWOG-S0600; SWOG-S0600; CDR0000551934; ECOG-SWOG-S0600; CAN-NCIC-SWOG-S0600; NCCTG-SWOG-S0600; S0600 (Other: Southwest Oncology Group); S0600 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-03

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil; Cetuximab; Bevacizumab

ARMS (3):
- Arm I (chemotherapy, cetuximab) (Experimental): Patients receive single-agent irinotecan hydrochloride IV or FOLFIRI IV. They also receive cetuximab IV over 1-2 hours on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab
- Arm II (chemotherapy, cetuximab, bevacizumab) (Experimental): Patients receive single-agent irinotecan hydrochloride or FOLFIRI AND cetuximab as in arm I. Patients also receive bevacizumab IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab; Biological: bevacizumab
- Arm III (closed to accrual as of 4/20/2009) (Experimental): Patients receive single-agent irinotecan hydrochloride or FOLFIRI AND cetuximab as in arm I. Patients also receive a higher dose of bevacizumab (higher than in arm II) IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab; Biological: bevacizumab

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm II (chemotherapy, cetuximab, bevacizumab); Arm III (closed to accrual as of 4/20/2009)

SUMMARY:
This randomized phase III trial is studying giving irinotecan and cetuximab together with bevacizumab to see how well it works compared with giving irinotecan and cetuximab alone in treating patients with metastatic colorectal cancer that progressed during first-line therapy. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether irinotecan and cetuximab are more effective with or without bevacizumab in treating metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare progression-free survival of patients with metastatic colorectal cancer that progressed on first-line therapy comprising bevacizumab and FOLFOX, OPTIMOX, or XELOX treated with irinotecan hydrochloride-based chemotherapy and cetuximab with vs without bevacizumab.

II. Compare overall survival of patients treated with these regimens. III. Compare objective tumor response (confirmed and unconfirmed, complete and partial response) in patients with measurable disease treated with these regimens.

IV. Compare the tolerability and safety profile of these regimens in these patients.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to Zubrod performance status (0 vs 1 or 2), discontinuation of oxaliplatin during first-line therapy (yes vs no), planned concurrent chemotherapy (FOLFIRI vs single-agent irinotecan hydrochloride), and time from last dose of bevacizumab (14-42 days vs >= 43 days).

All patients receive 1 of the following chemotherapy regimens:

SINGLE AGENT IRINOTECAN HYDROCHLORIDE: Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

FOLFIRI: Patients receive irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46-48 hours on days 1 and 2. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Patients are then randomized to 1 of 3 treatment arms.

ARM I: Patients receive single-agent irinotecan hydrochloride or FOLFIRI as outlined above and cetuximab IV over 1-2 hours on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive single-agent irinotecan hydrochloride or FOLFIRI as outlined above and cetuximab as in arm I. Patients also receive bevacizumab IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.

ARM III (closed to accrual as of 4/20/2009): Patients receive single-agent irinotecan hydrochloride or FOLFIRI as outlined above and cetuximab as in arm I. Patients also receive a higher dose of bevacizumab (higher than in arm II) IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 2 years and then once a year for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic colorectal cancer that has been histologically or cytologically confirmed; confirmation may be from either the primary tumor or a metastasis; patients must have wild type KRAS
* Patients must be registered within 28 days of documented disease progression on first line chemotherapy with bevacizumab plus either FOLFOX, OPTIMOX, or XELOX; this progression must have occurred within 90 days after the last dose of bevacizumab; patients who discontinued oxaliplatin, continued with 5-FU/LV or capecitabine and bevacizumab and then had subsequent progression while on fluoropyrimidine and bevacizumab are eligible; patients who discontinued bevacizumab due to adverse events in the first-line setting are not eligible
* Measurable or nonmeasurable disease
* At least 14 days must have elapsed since the last dose of first line chemotherapy and bevacizumab
* Patients must not have received prior treatment with irinotecan (either as adjuvant or metastatic treatment)
* Patients must have no history of prior treatment with cetuximab or other agents targeting VEGF or EGFR (except for bevacizumab)
* Prior radiotherapy is allowed, provided at least 28 days have elapsed since the last treatment; all adverse events related to radiation therapy must be resolved
* Prior surgery is allowed, provided at least 28 days have elapsed since any major surgery and patient has recovered from all effects
* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvate transaminase (SGPT) =< 2.5 x IULN; if there are known liver metastases, SGOT or SGPT must be =< 5 x IULN; these results must be obtained within 28 days prior to registration
* Serum creatinine =< IULN or measured or estimated creatinine clearance >= 60 mL/min
* Patients must not have a history or known presence of brain metastasis
* Patients may be on full dose anticoagulation with warfarin provided that the patient has an acceptable International Normalized Ratio (INR) (between 2 and 3), obtained within 28 days prior to registration
* No clinically relevant bleeding diathesis or coagulopathy
* Patients must not have experienced nephrotic range proteinuria from prior bevacizumab therapy; urine protein must be screened by urine analysis for Urine Protein Creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1,000 mg for patient enrollment; urine protein and creatinine used in calculating the UPC ratio must be obtained within 28 days prior to registration
* No uncontrolled high blood pressure (BP) (i.e., systolic BP > 150 mm Hg and diastolic BP > 90 mm Hg)
* No cardiovascular event within the past 6 months, including any of the following:

  * Arterial thrombosis
  * Unstable angina
  * Myocardial infarction
  * Cerebrovascular accident
* Patients must not have New York Heart Association (NYHA) >= Grade 2 congestive heart failure
* Patients must not have unstable symptomatic arrhythmia requiring medication; (patients with chronic, controlled arrhythmias such as atrial fibrillation or paroxysmal supraventricular tachycardia [PSVT] are eligible)
* No clinically significant peripheral vascular disease
* No serious or nonhealing active wound, ulcer, or bone fracture
* No history of gastrointestinal (GI) perforation while on prior bevacizumab
* No significant bleeding episodes (e.g., hemoptysis or upper or lower GI bleeding) within the past 6 months unless the source of bleeding has been resected
* No known hypersensitivity to bevacizumab or known potential hypersensitivity to cetuximab
* No other concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other type of anticancer treatment
* Due to the possibility of harm to a fetus or nursing infant from this treatment regimen, patients must not be pregnant or nursing; women and men of reproductive potential must have agreed to use an effective contraceptive method
* No other malignancy within the past 5 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gold, Principal Investigator — SWOG Cancer Research Network
Locations (382):
- United States (382):
  - Saint Edward Mercy Medical Center, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Medical Center, Duarte, California
  - Northbay Cancer Center, Fairfield, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin General Hospital, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - University of Southern California, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Palchak David MD, Pismo Beach, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Sutter Roseville Medical Center, Roseville, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Tahoe Forest Cancer Center, Truckee, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Bayhealth Medical Center at Kent General, Dover, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Edna Williams Cancer Center at the Baptist Cancer Institute, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Space Coast Cancer Centers-Titusville, Titusville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Memorial Hospital at Easton - Shore Regional Cancer Center, Easton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Montefiore Medical Center, The Bronx, New York
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Health Partners Regional Medical Center, Elyria, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Mansfield General Hospital-MedCentral Health System, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Bay Area Hospital, Coos Bay, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Riddle Hospital, Media, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Instutite/Greenville CCOP, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Tennessee - Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital - Luther Campus, Eau Claire, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Medical Consultants Limited, Milwaukee, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I: Chemotherapy + Cetuximab; Cohort II: Chemotherapy + Cetuximab: Single-agent irinotecan hydrochloride IV or FOLFIRI IV and cetuximab IV over 1-2 hours on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen)
- Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab: Single-agent irinotecan hydrochloride IV or FOLFIRI IV, cetuximab IV over 1-2 hours, and a lower dose of bevacizumab IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen)
- Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab: Single-agent irinotecan hydrochloride IV or FOLFIRI IV, cetuximab IV over 1-2 hours, and a higher dose of bevacizumab IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen)
- Cohort II: Chemotherapy + Bevacizumab: Single-agent irinotecan hydrochloride IV or FOLFIRI IV and a lower dose of bevacizumab IV over 30 minutes on day 1. Courses repeat every 14-21 days (depending upon chemotherapy regimen)
Period: Overall Study
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Started | 16 | 18 | 17 | 9 | 12
Eligible | 14 | 16 | 16 | 8 | 12
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 18 | 17 | 9 | 12
Not completed — Adverse Event | 2 | 2 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Progression | 10 | 12 | 9 | 6 | 10
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Not protocol specified | 2 | 0 | 3 | 1 | 0
Not completed — Ineligible | 2 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab | Total
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 12 | 66
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 76] | 63 [37 to 77] | 58 [46 to 75] | 65 [47 to 73] | 59 [38 to 70] | 60 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 2 | 7 | 28
  Male | 8 | 8 | 11 | 6 | 5 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 2 | 2 | 11
  Not Hispanic or Latino | 12 | 13 | 12 | 6 | 9 | 52
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 3
  White | 11 | 12 | 12 | 7 | 11 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 1 | 1 | 8
Performance Status [Number; unit: participants] — Patients graded according to the Zubrod Performance Status Scale: 0 is fully active, able to carry on all pre-disease performance without restriction; 1 is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 is ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours; 3 is capable of limited self-care, confined to bed or chair more than 50% of waking hours; and 4 is completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  participants
    0 | 9 | 8 | 8 | 1 | 4 | 30
    >= 1 | 5 | 8 | 8 | 7 | 8 | 36
Discontinuation of oxaliplatin while on first-line treatment [Number; unit: participants]
  Discontinued | 5 | 9 | 8 | 4 | 9 | 35
  Did not discontinue | 9 | 7 | 8 | 4 | 3 | 31
Planned concurrent chemotherapy [Number; unit: participants]
  FOLFIRI | 10 | 11 | 12 | 5 | 8 | 46
  Single-agent irinotecan | 4 | 5 | 4 | 3 | 4 | 20
Time from last dose of bevacizumab [Number; unit: participants]
  14-42 days | 12 | 13 | 13 | 6 | 8 | 52
  43 days or higher | 2 | 3 | 3 | 2 | 4 | 14

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: Time to death is from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 5 years
Population: No participants were analyzed due to limited accrual.
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Objective Tumor Response
Time Frame: Up to 5 years
Population: No participants were analyzed due to limited accrual.
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from date of registration to first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 5 years
Population: All eligible patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 12
months | 3.2 [1.4 to 3.8] | 4.2 [2.2 to 6.7] | 8.5 [2.2 to 9.4] | 1.4 [1.2 to 4.4] | 5.6 [3.4 to 6.9]

4. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3 through 5 adverse events that are related to study drug. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Number analyzed (Participants) | 14 | 16 | 16 | 7 | 12
Participants
  Albumin, serum-low (hypoalbuminemia) | 1 | 0 | 0 | 0 | 0
  Alkaline phosphatase | 0 | 0 | 1 | 1 | 0
  Anorexia | 0 | 1 | 0 | 0 | 1
  Bilirubin (hyperbilirubinemia) | 1 | 0 | 0 | 0 | 1
  Colitis, infectious (e.g., Clostridium difficile) | 0 | 0 | 1 | 0 | 0
  Confusion | 1 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 1
  Cough | 0 | 0 | 0 | 0 | 1
  Dehydration | 2 | 0 | 2 | 0 | 1
  Diarrhea | 3 | 2 | 3 | 3 | 5
  Dyspnea (shortness of breath) | 0 | 1 | 0 | 0 | 0
  Edema: limb | 0 | 0 | 1 | 0 | 0
  Edema: trunk/genital | 0 | 0 | 1 | 0 | 0
  Encephalopathy | 1 | 0 | 0 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 0 | 1 | 3 | 0 | 2
  Febrile neutropenia | 2 | 2 | 1 | 0 | 0
  Hemoglobin | 1 | 1 | 0 | 1 | 1
  Hemorrhage, GI - Stoma | 0 | 0 | 0 | 0 | 1
  Hypertension | 0 | 0 | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Abdomen NOS | 1 | 0 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1 | 0 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 0 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS | 0 | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1 | 0 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Mucosa | 0 | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 0 | 1 | 0 | 0 | 1
  Leukocytes (total WBC) | 5 | 4 | 2 | 2 | 0
  Lymphopenia | 0 | 0 | 1 | 0 | 0
  Magnesium, serum-low (hypomagnesemia) | 0 | 0 | 1 | 0 | 0
  Mental status | 1 | 0 | 0 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 0 | 1 | 1 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Oral cav | 0 | 0 | 1 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Pharynx | 0 | 0 | 0 | 0 | 1
  Nasal cavity/paranasal sinus reactions | 0 | 0 | 0 | 0 | 1
  Nausea | 0 | 1 | 3 | 0 | 0
  Neuropathy: sensory | 0 | 0 | 0 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 4 | 7 | 7 | 3 | 3
  Pain - Pain NOS | 0 | 0 | 0 | 0 | 1
  Phosphate, serum-low (hypophosphatemia) | 0 | 0 | 0 | 1 | 0
  Platelets | 1 | 2 | 0 | 0 | 0
  Pneumonitis/pulmonary infiltrates | 1 | 0 | 0 | 0 | 0
  Potassium, serum-low (hypokalemia) | 0 | 2 | 0 | 1 | 0
  Rash/desquamation | 0 | 1 | 1 | 0 | 0
  Rash: acne/acneiform | 3 | 2 | 4 | 2 | 0
  Rash: hand-foot skin reaction | 0 | 0 | 1 | 0 | 0
  Sodium, serum-low (hyponatremia) | 0 | 0 | 0 | 0 | 1
  Thrombosis/thrombus/embolism | 0 | 0 | 0 | 1 | 0
  Vomiting | 0 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Cohort I: Chemotherapy + Cetuximab | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab | Cohort II: Chemotherapy + Cetuximab | Cohort II: Chemotherapy + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 3/14 | 7/16 | 3/16 | 3/7 | 0/12
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16 | 15/16 | 7/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Chemotherapy + Cetuximab (N=14) | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab (N=16) | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab (N=16) | Cohort II: Chemotherapy + Cetuximab (N=7) | Cohort II: Chemotherapy + Bevacizumab (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0
Obstruction, GI - Ileum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 0 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection-Other (Specify) (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 0 | 1 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 0 | 1 | 0
Obstruction, GU - Bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Chemotherapy + Cetuximab (N=14) | Cohort I: Chemotherapy + Cetuximab + Lower Bevacizumab (N=16) | Cohort I: Chemotherapy + Cetuximab + Higher Bevacizumab (N=16) | Cohort II: Chemotherapy + Cetuximab (N=7) | Cohort II: Chemotherapy + Bevacizumab (N=12)
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 11 | 7 | 9 | 6 | 10
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
SVT and nodal arrhythmia - SVT arrhythmia NOS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Pain - External ear (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Dry eye syndrome (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular/Visual-Other (Specify) (Eye disorders) | 0 | 1 | 0 | 0 | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision-blurred vision (Eye disorders) | 1 | 2 | 2 | 1 | 0
Watery eye (epiphora, tearing) (Eye disorders) | 1 | 3 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 4 | 9 | 6 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 13 | 11 | 3 | 10
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Fistula, GI - Abdomen NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 1
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Incontinence, anal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3 | 6 | 7 | 2 | 2
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 3 | 3 | 8 | 3 | 4
Nausea (Gastrointestinal disorders) | 8 | 6 | 13 | 3 | 9
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 6 | 8 | 2 | 6
Pain - Anus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Pain - Rectum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7 | 8 | 1 | 8
Constitutional Symptoms-Other (Specify) (General disorders) | 0 | 1 | 0 | 0 | 0
Edema: limb (General disorders) | 4 | 0 | 3 | 1 | 2
Edema: trunk/genital (General disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 | 10 | 13 | 6 | 10
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2 | 1 | 1 | 1 | 1
Flu-like syndrome (General disorders) | 1 | 1 | 1 | 1 | 0
Injection site reaction/extravasation changes (General disorders) | 0 | 1 | 0 | 0 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 0 | 0 | 0 | 1
Pain - Pain NOS (General disorders) | 0 | 0 | 0 | 0 | 1
Pain-Other (Specify) (General disorders) | 0 | 0 | 0 | 0 | 1
Rigors/chills (General disorders) | 2 | 0 | 1 | 0 | 1
Pain - Liver (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Abdomen NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - UTI (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Mucosa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Muscle (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Pharynx (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Ungual (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection with unknown ANC - Conjunctiva (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection-Other (Specify) (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hemorrhage, GI - Stoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 | 3 | 3 | 2 | 2
AST, SGOT (Investigations) | 2 | 6 | 7 | 2 | 7
Alkaline phosphatase (Investigations) | 6 | 8 | 6 | 4 | 7
Bilirubin (hyperbilirubinemia) (Investigations) | 3 | 2 | 3 | 0 | 3
Creatinine (Investigations) | 2 | 1 | 0 | 0 | 4
INR (of prothrombin time) (Investigations) | 0 | 1 | 0 | 0 | 2
Leukocytes (total WBC) (Investigations) | 10 | 9 | 9 | 3 | 7
Lymphopenia (Investigations) | 1 | 1 | 1 | 1 | 2
Metabolic/Laboratory-Other (Specify) (Investigations) | 0 | 0 | 0 | 0 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 8 | 8 | 12 | 3 | 7
Platelets (Investigations) | 2 | 5 | 4 | 0 | 6
Weight loss (Investigations) | 1 | 3 | 5 | 3 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 | 8 | 4 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 3 | 4 | 8 | 2 | 8
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 | 4 | 5 | 3 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 | 4 | 8 | 3 | 8
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 | 6 | 9 | 3 | 5
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 | 6 | 6 | 4 | 5
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 | 1 | 3 | 3 | 7
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 5
Ataxia (incoordination) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 1 | 3
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Mental status (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Neuropathy: sensory (Nervous system disorders) | 2 | 7 | 5 | 4 | 6
Ocular/Visual-Other (Specify) (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 2
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 1 | 1 | 1 | 2 | 2
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 2 | 3
Mood alteration - anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 0 | 2 | 2 | 1
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pain - Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 5 | 4 | 0 | 5
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1
Urine color change (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4 | 1 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 1
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 2 | 5
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Mucositis/stomatitis (functional/symp) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7 | 4 | 3 | 1
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 | 4 | 5 | 3 | 7
Nail changes (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 3 | 0
Pain - Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 3 | 6 | 1 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 10 | 13 | 13 | 6 | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hot flashes/flushes (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Due to inadequate accrual, study was terminated and limited outcome data was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less